CLINICAL TRIAL: NCT03468790
Title: A Multi-centre, Randomized, Double-blind, Placebo-controlled Phase III Study to Evaluate the Efficacy and Safety of Anti-IgE Monoclonal Antibody to Treat Allergic Asthma Patients Not Adequately Controlled Despite Med/High ICS/LABA.
Brief Title: Anti-IgE Monoclonal Antibody Treatment in Patients With Allergic Asthma.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Biomabs Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C007AAIII
Record Dates: First submitted 2018-03-07; First posted 2018-03-19 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2020-03

CONDITIONS: Asthma, Allergic
MeSH Terms: conditions — Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination; Budesonide; Inhalation; Fluticasone-Salmeterol Drug Combination; Albuterol

STUDY DESIGN:
Intervention Model Description: placebo parallel-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CMAB007 + Seretide/Symbicort + Ventolin (Experimental): CMAB007(recombinant humanized anti-IgE monoclonal antibody for injection ) will be at a fixed dose determined by the subjects' total IgE and weight at V0. All the subjects will be treated subcutaneously for 24 weeks. The 4-week total dose is 0.016mg/kg/IgE(IU/ml), administered every 2 or 4 weeks, for the subjects with total IgE level 60-700IU/ml. If the total IgE level is 700-1500IU/ml, they will be administered 375mg every 2 weeks. Symbicort(Budesonide and formoterol fumarate powder for inhalation) or Seretide (salmeterol xinafoate and fluticasone propionate powder for inhalation) will be used 1/2 inhalations bid as asthma-controlled drug during the whole study. Ventolin (Salbutamol sulphate aerosol) will be used as asthma rescue drug.
  Interventions: Drug: CMAB007; Drug: Symbicort; Drug: Seretide; Drug: Ventolin
- Placebo + Seretide/Symbicort + Ventolin (Placebo Comparator): Placebo is without active components of the study drug and used as same as the study drug.
  Interventions: Drug: Symbicort; Drug: Seretide; Drug: Ventolin; Drug: placebo

INTERVENTIONS:
Drug: CMAB007 — the study drug
  Other Names: recombinant humanized anti-IgE monoclonal antibody
  Arms: CMAB007 + Seretide/Symbicort + Ventolin
Drug: Symbicort — asthma-controlled drug
  Other Names: budesonide and formoterol fumarate powder for inhalation
Drug: Seretide — asthma-controlled drug
  Other Names: salmeterol xinafoate and fluticasone propionate
Drug: Ventolin — asthma rescue drug
  Other Names: Salbutamol sulphate aerosol
Drug: placebo — No active components
  Arms: Placebo + Seretide/Symbicort + Ventolin

SUMMARY:
This is a multi-centre, randomized, double-blind，placebo parallel-controlled phase III study to evaluate the efficacy and safety of CMAB007 (recombinant humanized anti-immunoglobulin E(IgE) monoclonal antibody for injection) to treat asthma patients who remain not adequately controlled despite Med/high ICS plus LABA in China. Following a screening period of up to 2 weeks and run-in period of 4 weeks, randomized patients will enter a 24-week treatment period with CMAB007 or placebo. Efficacy and safety will be assessed at 4-week intervals during the treatment period.

DETAILED DESCRIPTION:
Approximately 400 asthma patients with an increased serum total IgE level(60-1500 international unit(IU)/ml) and uncontrolled receiving medium to high dose inhaled corticosteroid (ICS) plus long-acting β2-agonist(LABA) will be randomised in about 43 sites in China. They will be administered CMAB007 or placebo at a ratio of 2:1 for 24 weeks. During the whole study, all subjects will be on regularly fixed combination of med/high ICS and LABA (budesonide and formoterol fumarate powder for inhalation or salmeterol xinafoate and fluticasone propionate powder for inhalation). They should complete PEF measurement and patient diary daily and be assessed every 4 weeks. Spirometry, questionnaires, laboratory tests and so on will be performed. At selected sites, about 45 patients will be enrolled in a sub-study to assess the pharmacokinetic and pharmacodynamic characterises of CMAB007. Anti-drug antibody (ADA) will be sampled at V1, V2 and V7 too.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent prior to any study assessment;
2. Age 15-75 years inclusive, female or male;
3. Diagnosed as asthma according to the guideline for the prevention and treatment of bronchial asthma in China (version 2016), with duration for more than 1 years;
4. Have had at least one severe asthma exacerbations(requiring systemic steroid use) in the previous one year;
5. At screening, serum total IgE level 60-1500IU/ml and body weight 20-150kg.
6. Receiving seretide(fluticasone>250ug/day) or symbicort(budesonide>400ug/day) for at least 3 months and stable dose for at least 4 weeks prior to screening. Asthma symptom control level is still partly controlled or uncontrolled. Detailed drugs and usage are one of the following: Seretide 50/250ug 1 inhalation bid；Seretide 50/500ug 1 inhalation bid；Symbicort 160/4.5ug 2 inhalations bid or Symbicort 320/9ug 1 inhalation bid.
7. None of other asthma controller medications other than seretide or symbicort including systemic steroid, leukotriene modifiers, theophylline, histamine1 receptor blockers, anticholinergic drugs, traditional Chinese medicine and so on have been used 2 weeks prior to screening.
8. At screening, FEV1 < 80% of the predicted normal value.
9. At screening, laboratory tests results should meet all of the following: hemoglobin≥80g/l；3*10^9/l≤white blood cell≤10*10^9/l；platelet≥75*10^9/l；liver function(glutamic-pyruvic transaminase, glutamic-oxalacetic transaminase and total bilirubin)≤2*upper limit of normal value；renal function≤1.5*upper limit of normal value.
10. At screening, pregnant test is negative,or not lactating, for women of child-bearing potential. Effective methods of contraception will be maintained throughout the study and 6 months after the study.
11. Can understand and complete questionnaires correctly, complete PEF and patient diary correctly, and be followed up according to scheduled table.

Exclusion Criteria:

1. History of critical asthma exacerbations，such as tracheal intubation or intensive care unit admission.
2. Currently smoker, or a former smoker with a smoking history > 10 pack-years(defined as the number of packs of 20 cigarettes smoked per day multiplied by number of years the patient smoked).
3. Have elevated serum IgE levels for other causes other than allergens, such as parasite infections, allergic bronchopulmonary aspergillosis, Churg-Strauss syndrome and so on.
4. Desensitization therapy or immunosuppressant agents such as cyclosporine, methotrexate and gold preparation during 3 months prior to screening.
5. Biological agents such as monoclonal antibody including investigational biological drugs during 6 months prior to screening.
6. Vaccinated live/attenuated virus or bacterial vaccines, or intravenous used immunoglobulin G, during 4 weeks prior to screening.
7. History of bronchial thermoplasty for asthma during 12 months prior to screening.
8. Use of any anti-IgE monoclonal antibody including Xolair for asthma during 12 months prior to screening.
9. Respiratory infections（such as pneumonia,upper respiratory tract infection，etc）or large surgeries during 4 weeks prior to screening.
10. Combined with other pulmonary diseases, such as chronic obstructive pulmonary disease, bronchiectasis, pulmonary interstitial fibrosis, etc.
11. History of malignancies other than squamous cell carcinoma or basal cell carcinoma of the skin and carcinoma in situs of cervix with complete excision and no evidence of recurrences.
12. Acquired immune deficiency syndrome or human immunodeficiency virus infection patients.
13. History of malignant or proliferative diseases of the lymphatic system such as lymphoma, or there are symptoms and signs indicating lymphatic proliferative diseases, or splenomegaly (≥2cm under the ribs).
14. With uncontrolled hypertension(systolic pressure ≥160 or diastolic pressure ≥100 in millimeters of mercury) at screening.
15. With severe, progressive or uncontrolled hepatic, renal, gastrointestinal, cardio-cerebral vascular, hematopoietic，genitourinary, endocrine, nervous and immunological medical conditions, or other conditions that investigators think the patient not suitable for this study.
16. Have a history of drug or alcohol abuse or poor compliance of drugs.
17. With known hypersensitivity to human immunoglobulin, anti-IgE monoclonal antibody for injection or components.
18. Have attended other clinical trials of investigational drugs, or within 30 days or 5 half-lives of enrollment, whichever is longer.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 393 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-03-09 (Actual)

PRIMARY OUTCOMES:
the mean number of asthma exacerbations per patient during the 24-week treatment period | from baseline(0 week) to 24 weeks
  Asthma exacerbation is defined by a worsening of asthma symptoms resulting in: 1.out-planned outpatient visit; 2.use of systemic and/or nebulized inhaled corticosteroids; 3.emergency room visit; 4. hospitalization.

SECONDARY OUTCOMES:
the proportion of patients with asthma exacerbations during the 24-week treatment period | from baseline(0 week) to 24 weeks
  the number of patients with at least one exacerbations divided by the total number of patients.
time to the first asthma exacerbation during treatment period | from baseline(0 week) to 24 weeks
  the time from baseline to the first asthma exacerbation
change from baseline in asthma symptom scores(daytime, nocturnal and total) over the 24-week treatment period | from baseline(0 week) to 24 weeks
  mean asthma symptom scores(daytime, nocturnal and total): (pre-treatment - post-treatment)/pre-treatment *100%
change from baseline in Asthma Control Test(ACT) over the 24-week treatment period | from baseline(0 week) to 24 weeks
  ACT total score: (pre-treatment - post-treatment)/pre-treatment *100%
change from baseline in Asthma Quality of Life Questionnaire(AQLQ) over the 24-week treatment period | from baseline(0 week) to 24 weeks
  AQLQ total score and threshold score: (pre-treatment - post-treatment)/pre-treatment *100%
investigator's and patient's Global Evaluation of Treatment Effectiveness(GETE) over 16 and 24-week treatment period | from baseline(0 week) to 16 and 24 weeks
  GETE score at week 16 and 24
change from baseline in rescue medication use over the 24-week treatment period | from baseline(0 week) to 24 weeks
  mean rescue medication use(puff/day): (pre-treatment - post-treatment)/pre-treatment *100%
change from baseline in lung function parameters(FEV1,FVC and FEV1/FVC) over the 24-week treatment period | from baseline(0 week) to 24 weeks
  FEV1,FVC and FEV1/FVC values: (post-treatment - pre-treatment)/pre-treatment *100%
change from baseline in mean peak expiratory flow(PEF) over the 24-week treatment period | from baseline(0 week) to 24 weeks
  mean PEF value: (post-treatment - pre-treatment)/pre-treatment *100%

CONTACTS AND LOCATIONS:
Overall Officials: Nanshan Zhong, M.D., Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (2):
- China (2):
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lai K, Yan Z, Qian D, Zhang X, Bian T, Dai X, Li H, Lin L, Wang J, Wang L, Yang J, Hu Y, Li H, Nie X, Jin F, Li G, Sun S, Xu F, Zhao H, Chen Y, Liu C, Zhu H, Li J, Guo Y, Zhong N. Benefits of CMAB007 in Chinese Patients Having Inadequately Controlled Moderate/Severe Asthma With Increased Total IgE: A Randomized Phase 3 Trial. Allergy Asthma Immunol Res. 2026 Jan;18(1):39-54. doi: 10.4168/aair.2026.18.1.39. Epub 2025 Nov 26. PMID 41345745